CLINICAL TRIAL: NCT00172211
Title: Comparison of Oxidative Stress and Insulin Resistance Before and After Using Physioneal in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Shao-Yu Yang, Attending Physician, Nation Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 185-CL4
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2007-01

CONDITIONS: Kidney Failure,Chronic
Keywords: Physioneal; Peritoneal dialysis; Oxidative stress; insulin resistance
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance

INTERVENTIONS:
Drug: Physioneal

SUMMARY:
Patients affected by end-stage renal disease (ESRD) are subjected to enhanced oxidative stress, as a result of reduced anti-oxidant systems and increased pro-oxidant activity. Besides, insulin resistance is also very common in ESRD patients. Both enhanced oxidative stress and insulin resistance increase the risk of atherosclerosis and cardiovascular mortality, and intention to reduce oxidative stress and insulin resistance is important in ESRD patients who suffer from high cardiovascular risk.

The high concentration of glucose and glucose degradation products (GDP), high lactate, and low pH in conventional peritoneal dialysis (PD) solutions are known as bioincompatible factors, which are believed to increase oxidative stress in PD patients. Physioneal®, a more biocompatible dialysis solution with neutral pH, physiologic bicarbonate concentration and low GDP level, has been applied in Europe for several years. Previous studies of Physioneal® have revealed advantages of improved infusion pain, more efficient acid-base control, increased ultrafiltration, and reduced peritonitis duration. However, its effects on oxidative stress and insulin resistance in peritoneal dialysis patients are not reported yet. The comparison of oxidative stress and insulin resistance before and after using Physioneal® may help to elucidate the possibly beneficial effects on uremic patients, which frequently suffer from increased oxidative stress and insulin resistance.

Thirty continuous ambulatory peritoneal dialysis (CAPD) patients will be selected in this study, and receive conventional solution (Dianeal® PD-2 or PD-4) for a baseline period of 3 months. Then Physioneal® will be used for 3 months. Clinical conditions, biochemical and hematological parameters, oxidative markers in blood and effluent, and insulin resistance will be measured at baseline, before and after Physioneal®, and some markers will be measured 1 month after discontinuing Physioneal® and changing back to conventional solution. The medication used in each patient will be recorded, and the dialysis prescription will be adjusted by a nephrologist according to clinical data. The data collected before and after Physioneal® will be analyzed by paired-t test.

DETAILED DESCRIPTION:
Patients affected by end-stage renal disease (ESRD) are subjected to enhanced oxidative stress, as a result of reduced anti-oxidant systems and increased pro-oxidant activity. Enhanced oxidative stress in uremic patients increases the risk of atherosclerosis and cardiovascular mortality. Furthermore, bioincompatibility of dialysis therapy further increases oxidative stress. High concentration of glucose, high lactate, low pH, and/or high concentration of glucose degradation products (GDP) are known as bioincompatible factors and believed to increase oxidative stress in peritoneal dialysis patients. A more biocompatible dialysis solution, i.e., neutral pH, containing physiologic concentration of bicarbonate and low concentration of GDP has been developed. There is a growing body of in vitro studies showing this neutral bicarbonate containing dialysis solution more biocompatible compared to conventional solutions. However, its effects on oxidative stress in peritoneal dialysis patients are not reported yet. On the other hand, insulin resistance is associated with cardiovascular disease, and it is very common in uremic patients. Some animal studies suggested that reduced oxidative stress enhanced insulin sensitivity, and the effects of reduced oxidative stress in human have not been extensively investigated. Previous studies of Physioneal®, a kind of more biocompatible dialysis solution which contains bicarbonate, have revealed advantages of improved infusion pain, more efficient acid-base control, increased ultrafiltration, and reduced peritonitis duration. The comparison of oxidative stress and insulin resistance before and after using Physioneal®, may help to elucidate the possibly beneficial effects on uremic patients, which frequently suffer from increased oxidative stress and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old, younger than 70 years old
2. Non-diabetic ESRD patients, e.g. chronic glomerulonephritis, hypertensive nephrosclerosis, interstitial nephritis, polycystic kidney disease, etc.
3. Undergoing CAPD for at least 3 months and less than 60 months
4. Kt/Vurea (normalized by Watson's method) is greater than 1.7, and serum albumin is greater than 3.5 g/dL

Exclusion Criteria:

1. Unstable clinical conditions or evidence of malignancy
2. Diabetes mellitus
3. Pregnancy
4. Have peritonitis in recent 3 months or other active bacterial infections
5. Taking any medication known to markedly interfere oxidative stress, e.g. large dose of vitamin C (greater than 500 mg/day) or vitamin E (greater than 400 IU/day).
6. Medical history of systemic lupus erythematosus or rheumatoid arthritis
7. Serum potassium is less than 3.0 mEq/l
8. Participate in another study that would interfere with the outcome of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The oxidative markers in month 3, 6, and 7
The insulin resistance in month 3, 6, and 7

SECONDARY OUTCOMES:
The hematologic, biochemical markers, and peritoneal function
in month 3,6, and 7

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, Ph.D. & M.D., Principal Investigator — Section of Nephrology, Department of Internal Medicine, National Taiwan University
Locations (1):
- Taiwan Universithy Hospital, Taipei, Taiwan